CLINICAL TRIAL: NCT01328028
Title: Hospital-based Epidemiological Study on the Distribution of Human Papillomavirus (HPV) Types in Adult Women Diagnosed With Invasive Cervical Cancer (ICC) in New Zealand
Brief Title: Human Papillomavirus (HPV) Type Distribution in Adult Women Diagnosed With Invasive Cervical Cancer in New Zealand
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111050
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2011-06

CONDITIONS: Cervical Cancer
Keywords: Invasive cervical cancer; Human papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cervical specimen

GROUPS / COHORTS (1):
- Group A: Subjects diagnosed with invasive cervical cancer
  Interventions: Other: Testing of archived cervical cancer tissue samples; Other: Data collection

INTERVENTIONS:
Other: Testing of archived cervical cancer tissue samples — Cervical samples will be tested for histopathology diagnosis and human papillomavirus deoxyribonucleic acid testing.
Other: Data collection — Log sheet

SUMMARY:
The aim of this study is to assess the distribution of the most frequent types of human papillomavirus in women diagnosed with invasive cervical cancer in New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* A female aged 18 years and above at the time of cervical specimen collection, and currently residing in New Zealand.
* Histological diagnoses of invasive cervical cancer stage IB or greater, within at least the last 3 years.
* Written informed consent obtained from the subject/ next of kin/ Legally acceptable representative.
* Availability of cervical specimen on which the diagnosis was made prior to any chemotherapy or radiotherapy.
* The cervical specimen should be of appropriate size and with regular tissue specimens.
* The cervical specimen should be adequately preserved.
* All links to the subject's identity should be removed from the paraffin block.

Exclusion Criteria:

Not Applicable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged >= 18 years at the time that the cervical specimen was taken, and diagnosed with invasive cervical cancer stage IB or greater
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of HPV-16 and HPV-18 in women with invasive cervical cancer | At least the last 3 years from the time of study start

SECONDARY OUTCOMES:
Occurrence of other high-risk HPV types in women with invasive cervical cancer | At least the last 3 years from the time of study start
Occurrence of HPV-16/ HPV-18 co-infection with other high-risk HPV types in women with invasive cervical cancer | At least the last 3 years from the time of study start
Occurrence of low-risk HPV types in women diagnosed with invasive cervical cancer | At least the last 3 years from the time of study start

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Sykes P, Gopala K, Tan AL, Kenwright D, Petrich S, Molijn A, Chen J. Type distribution of human papillomavirus among adult women diagnosed with invasive cervical cancer (stage 1b or higher) in New Zealand. BMC Infect Dis. 2014 Jul 8;14:374. doi: 10.1186/1471-2334-14-374. PMID 25000939